CLINICAL TRIAL: NCT00555906
Title: Phase 1/2 Open-label Study Of The Safety And Efficacy Of Pd 0332991 In Combination With Bortezomib And Dexamethasone In Patients With Refractory Multiple Myeloma
Brief Title: An Investigational Drug, Palbociclib (PD-0332991), Is Being Studied In Combination With Velcade And Dexamethasone In Patients With Multiple Myeloma. Patients Must Have Received Prior Treatment For Multiple Myeloma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5481004; 2010-022515-20 (EudraCT Number)
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Results first posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: PD 0332991

INTERVENTIONS:
Drug: Bortezomib — Escalating doses of bortezomib will be administered intravenously on Days 8, 11, 15 and 18 of a 28-day cycle (Schedule A) or of a 21-day cycle (Schedule B). The planned doses to be evaluated are 0.7, 1 and 1.3 mg/m2 in combination with PD 0332991 and dexamethasone.
  Other Names: Velcade
Drug: Dexamethasone — 20 mg, orally on Days 8, 11, 15 and 18 of a 28 day cycle (Schedule A) or of a 21-day cycle (Schedule B) in combination with PD 0332991 and bortezomib.
Drug: PD 0332991 — Escalating doses of PD 0332991 will be administered orally on Days 1-21 of a 28-day cycle for Schedule A and on Days 1-12 of a 21-day cycle for Schedule B. The planned doses to be evaluated are 50, 75, 100 mg and 125 mg once daily in combination with bortezomib and dexamethasone.

SUMMARY:
This is a Phase 1/2 study evaluating the safety and anti-tumor activity of PD 0332991 in combination with Velcade® [bortezomib] and dexamethasone in patients who have received at least one previous treatment for multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of symptomatic multiple myeloma as defined by International Myeloma Working Group (IMWGURC).
* Phase 1: Relapsed or relapsed/refractory myeloma after at least 1 previous treatments and with a life expectancy of more than 3 months.
* Phase 2: Measurable (as defined by IMWGURC) disease after at least 1 previous treatment.

Exclusion Criteria:

* History of allogeneic stem cell transplant.
* Phase 2 only: Prior bortezomib therapy will only be allowed if there was a demonstrated positive response, and disease progression occurred off therapy.
* Must have not experienced significant blood level changes, e.g. very low platelets, while on previous bortezomib therapy
* Prior radiation therapy to > 25% of the bone marrow (whole pelvis is 25%).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-01; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (15):
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Northwestern Memorial Hospital/Main Labs, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - University of Maryland, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Presbyterian, Weill Cornell Medical College, New York, New York
  - University of Pennsylvania Abramson Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
- Vseobecna fakultni nemocnice v Praze, Prague, Czechia
- Germany (2):
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Klinikum Johannes-Gutenberg -Universitaet, III. Medizinische Klinik und Poliklinik, Mainz

REFERENCES:
- [Derived] Niesvizky R, Badros AZ, Costa LJ, Ely SA, Singhal SB, Stadtmauer EA, Haideri NA, Yacoub A, Hess G, Lentzsch S, Spicka I, Chanan-Khan AA, Raab MS, Tarantolo S, Vij R, Zonder JA, Huang X, Jayabalan D, Di Liberto M, Huang X, Jiang Y, Kim ST, Randolph S, Chen-Kiang S. Phase 1/2 study of cyclin-dependent kinase (CDK)4/6 inhibitor palbociclib (PD-0332991) with bortezomib and dexamethasone in relapsed/refractory multiple myeloma. Leuk Lymphoma. 2015;56(12):3320-8. doi: 10.3109/10428194.2015.1030641. Epub 2015 May 15. PMID 25813205
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481004&StudyName=An%20Investigational%20Drug%2C%20Palbociclib%20%28PD-0332991%29%2C%20Is%20Being%20Studied%20In%20Combination%20With%20Velcade%20And%20Dexamethasone%20In%20Patients%20With%20M

RESULTS

PARTICIPANT FLOW:
Groups:
- Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule A): Palbociclib (PD 0332991) 100 milligram (mg) capsule orally once daily for 21 days followed by 7 days off-treatment in a 28-day cycle along with bortezomib 1.0 milligram per square meter (mg/m^2) intravenous injection and dexamethasone 20 mg tablet orally 30 minutes prior to bortezomib injection on Day 8, 11, 15 and 18 of 28-day cycle (schedule A) during Phase 1 of the study. Treatment was continued until any of the following withdrawal criteria was met: disease progression (unless the investigator judged that participant could still derive clinical benefit from continuing the treatment and the risk/benefit was still favorable), unacceptable toxicities, need for surgery or radiation therapy considered due to progressive disease by investigator, investigator conclusion that it is in the participant's best interest to discontinue therapy, need for anti-cancer therapy, lost to follow-up, withdrawal from treatment, or withdrawal of consent.
- Palbociclib 75mg+Bortezomib+Dexamethasone(Phase1:Schedule A): Palbociclib (PD 0332991) 75 mg capsule orally once daily for 21 days followed by 7 days off-treatment in a 28-day cycle along with bortezomib 1.0 mg/m^2 intravenous injection and dexamethasone 20 mg tablet orally 30 minutes prior to bortezomib injection on Day 8, 11, 15 and 18 of 28-day cycle (schedule A) during Phase 1 of the study. Treatment was continued until any of the following withdrawal criteria was met: disease progression (unless the investigator judged that participant could still derive clinical benefit from continuing the treatment and the risk/benefit was still favorable), unacceptable toxicities, need for surgery or radiation therapy considered due to progressive disease by investigator, investigator conclusion that it is in the participant's best interest to discontinue therapy, need for anti-cancer therapy, lost to follow-up, withdrawal from treatment, or withdrawal of consent.
- Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule B): Palbociclib (PD 0332991) 100 mg capsule orally once daily for 12 days followed by 9 days off-treatment in a 21-day cycle along with bortezomib 1.0 mg/m^2 intravenous injection and dexamethasone 20 mg tablet orally 30 minutes prior to bortezomib injection on Day 8, 11, 15 and 18 of 21-day cycle (schedule B) during Phase 1 of the study. Treatment was continued until any of the following withdrawal criteria was met: disease progression (unless the investigator judged that participant could still derive clinical benefit from continuing the treatment and the risk/benefit was still favorable), unacceptable toxicities, need for surgery or radiation therapy considered due to progressive disease by investigator, investigator conclusion that it is in the participant's best interest to discontinue therapy, need for anti-cancer therapy, lost to follow-up, withdrawal from treatment, or withdrawal of consent.
- Palbociclib 125mg+Bortezomib+Dexamethasone(Phase1:Schedule B): Palbociclib (PD 0332991) 125 mg capsule orally once daily for 12 days followed by 9 days off-treatment in a 21-day cycle along with bortezomib 1.0 mg/m^2 intravenous injection and dexamethasone 20 mg tablet orally 30 minutes prior to bortezomib injection on Day 8, 11, 15 and 18 of 21-day cycle (schedule B) during Phase 1 of the study. Treatment was continued until any of the following withdrawal criteria was met: disease progression (unless the investigator judged that participant could still derive clinical benefit from continuing the treatment and the risk/benefit was still favorable), unacceptable toxicities, need for surgery or radiation therapy considered due to progressive disease by investigator, investigator conclusion that it is in the participant's best interest to discontinue therapy, need for anti-cancer therapy, lost to follow-up, withdrawal from treatment, or withdrawal of consent.
- Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:ScheduleB): Palbociclib (PD 0332991) 100 mg capsule orally once daily for 12 days followed by 9 days off-treatment in a 21-day cycle along with bortezomib 1.0 mg/m^2 intravenous injection and dexamethasone 20 mg tablet orally 30 minutes prior to bortezomib injection on Day 8, 11, 15 and 18 of 21-day cycle (schedule B) during Phase 2 of the study. Treatment was continued until any of the following withdrawal criteria was met: disease progression (unless the investigator judged that participant could still derive clinical benefit from continuing the treatment and the risk/benefit was still favorable), unacceptable toxicities, need for surgery or radiation therapy considered due to progressive disease by investigator, investigator conclusion that it is in the participant's best interest to discontinue therapy, need for anti-cancer therapy, lost to follow-up, withdrawal from treatment, or withdrawal of consent.
Period: Phase 1
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule A) | Palbociclib 75mg+Bortezomib+Dexamethasone(Phase1:Schedule A) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule B) | Palbociclib 125mg+Bortezomib+Dexamethasone(Phase1:Schedule B) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:ScheduleB)
Started | 3 | 6 | 7 | 5 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 7 | 5 | 0
Not completed — Objective Progression or Relapse | 3 | 5 | 3 | 1 | 0
Not completed — Global Deterioration of Health Status | 0 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Period: Phase 2
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule A) | Palbociclib 75mg+Bortezomib+Dexamethasone(Phase1:Schedule A) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule B) | Palbociclib 125mg+Bortezomib+Dexamethasone(Phase1:Schedule B) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:ScheduleB)
Started | 0 | 0 | 0 | 0 | 32
Treated | 0 | 0 | 0 | 0 | 30
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 32
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 4
Not completed — Global Deterioration of Health Status | 0 | 0 | 0 | 0 | 2
Not completed — Objective Progression or Relapse | 0 | 0 | 0 | 0 | 16
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2
Not completed — Other | 0 | 0 | 0 | 0 | 6
Not completed — Randomized but not Treated | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all enrolled participants.
Groups:
- Palbociclib + Bortezomib + Dexamethasone (Phase1:Schedule A): Included all participants who received palbociclib (PD 0332991) 75 mg or 100 mg capsule orally once daily for 21 days followed by 7 days off-treatment in a 28-day cycle along with bortezomib 1.0 mg/m^2 intravenous injection and dexamethasone 20 mg tablet orally 30 minutes prior to bortezomib injection on Day 8, 11, 15 and 18 of 28-day cycle (schedule A) during Phase 1 of the study. Treatment was continued until any of the following withdrawal criteria was met: disease progression (unless the investigator judged that participant could still derive clinical benefit from continuing the treatment and the risk/benefit was still favorable), unacceptable toxicities, need for surgery or radiation therapy considered due to progressive disease by investigator, investigator conclusion that it is in the participant's best interest to discontinue therapy, need for anti-cancer therapy, lost to follow-up, withdrawal from treatment, or withdrawal of consent.
- Palbociclib + Bortezomib + Dexamethasone (Phase1:Schedule B): Included all participants who received palbociclib (PD 0332991) 100 mg or 125 mg capsule orally once daily for 12 days followed by 9 days off-treatment in a 21-day cycle along with bortezomib 1.0 mg/m^2 intravenous injection and dexamethasone 20 mg tablet orally 30 minutes prior to bortezomib injection on Day 8, 11, 15 and 18 of 21-day cycle (schedule B) during Phase 1 of the study. Treatment was continued until any of the following withdrawal criteria was met: disease progression (unless the investigator judged that participant could still derive clinical benefit from continuing the treatment and the risk/benefit was still favorable), unacceptable toxicities, need for surgery or radiation therapy considered due to progressive disease by investigator, investigator conclusion that it is in the participant's best interest to discontinue therapy, need for anti-cancer therapy, lost to follow-up, withdrawal from treatment, or withdrawal of consent.
- Palbociclib + Bortezomib + Dexamethasone (Phase2:ScheduleB): Included all participants who received palbociclib (PD 0332991) 100 mg capsule orally once daily for 12 days followed by 9 days off-treatment in a 21-day cycle along with bortezomib 1.0 mg/m^2 intravenous injection and dexamethasone 20 mg tablet orally 30 minutes prior to bortezomib injection on Day 8, 11, 15 and 18 of 21-day cycle (schedule B) during Phase 2 of the study. Treatment was continued until any of the following withdrawal criteria was met: disease progression (unless the investigator judged that participant could still derive clinical benefit from continuing the treatment and the risk/benefit was still favorable), unacceptable toxicities, need for surgery or radiation therapy considered due to progressive disease by investigator, investigator conclusion that it is in the participant's best interest to discontinue therapy, need for anti-cancer therapy, lost to follow-up, withdrawal from treatment, or withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Palbociclib + Bortezomib + Dexamethasone (Phase1:Schedule A) | Palbociclib + Bortezomib + Dexamethasone (Phase1:Schedule B) | Palbociclib + Bortezomib + Dexamethasone (Phase2:ScheduleB) | Total
Number analyzed (Participants) | 9 | 12 | 32 | 53
Age, Customized [Number; unit: participants]
  18 to 44 years | 2 | 1 | 0 | 3
  45 to 64 years | 4 | 7 | 13 | 24
  Greater than or equal to (>=) 65 years | 3 | 4 | 19 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 17 | 23
  Male | 4 | 11 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of PD-0332991: Phase 1
Description: MTD=highest dose level for which no more than 1 out of 6 participants experienced dose-limiting toxicity (DLT). DLT=any of the following treatment-related events: Absolute neutrophil count (ANC) less than (<)1000/microliter (mcL) (Grade 3 neutropenia) associated with documented infection/fever >=38.5degrees Celsius (C); Grade >=3 nonhematologic treatment-related toxicity, except those that were not maximally treated or considered tolerable, Grade 3 corrected QT interval (QTc) prolongation (QTc >500 millisecond [msec]) in asymptomatic participants even after repeat testing to exclude confounding factors and correction of reversible causes; Delay in the administration of Cycle 2 for more than 1 week of the planned date due to platelet count <25,000/mcL and/or ANC <500/mcL, or due to prolonged nonhematologic toxicities of Grade >=3; Inability to deliver at least 80 percent (%) of the planned PD 0332991 or bortezomib doses during Cycle 1 due to toxicity.
Time Frame: Day 1 up to Day 28 during Cycle 1 in schedule A, Day 1 up to Day 21 during Cycle 1 in schedule B
Population: DLT analysis set included all enrolled participants who received at least one dose of study treatment and did not have a major deviation in the first cycle.
Measure: Number; unit: milligram (mg)
Groups:
- Palbociclib + Bortezomib + Dexamethasone (Phase1:ScheduleB): Included all participants who received palbociclib (PD 0332991) 100 mg or 125 mg capsule orally once daily for 12 days followed by 9 days off-treatment in a 21-day cycle along with bortezomib 1.0 mg/m^2 intravenous injection and dexamethasone 20 mg tablet orally 30 minutes prior to bortezomib injection on Day 8, 11, 15 and 18 of 21-day cycle (schedule B) during Phase 1 of the study. Treatment was continued until any of the following withdrawal criteria was met: disease progression (unless the investigator judged that participant could still derive clinical benefit from continuing the treatment and the risk/benefit was still favorable), unacceptable toxicities, need for surgery or radiation therapy considered due to progressive disease by investigator, investigator conclusion that it is in the participant's best interest to discontinue therapy, need for anti-cancer therapy, lost to follow-up, withdrawal from treatment, or withdrawal of consent.
Arm/Group | Palbociclib + Bortezomib + Dexamethasone (Phase1:Schedule A) | Palbociclib + Bortezomib + Dexamethasone (Phase1:ScheduleB)
Number analyzed (Participants) | 9 | 12
milligram (mg) | NA — For Palbociclib + Bortezomib + Dexamethasone (Phase1:Schedule A), reported DLTs were >1/6 (exceeding the MTD criteria), hence no MTD could be determined for Schedule A. | 100

2. Primary Outcome: Recommended Phase II Dose (RP2D) of PD-0332991: Phase 1
Description: RP2D was determined based on the MTD, safety and tolerability profile of the study treatment.
Time Frame: Day 1 up to Day 28 during Cycle 1 in schedule A, Day 1 up to Day 21 during Cycle 1 in schedule B
Population: as for outcome 1
Measure: Number; unit: milligram (mg)
Arm/Group | Palbociclib + Bortezomib + Dexamethasone (Phase1:Schedule A) | Palbociclib + Bortezomib + Dexamethasone (Phase1:ScheduleB)
Number analyzed (Participants) | 9 | 12
milligram (mg) | NA — Both palbociclib 75 mg+bortezomib+dexamethasone and palbociclib 100 mg+bortezomib+dexamethasone had DLT >1/6, hence no RP2D was selected from these 2 dosing groups. | 100

3. Primary Outcome: Percentage of Participants With Objective Response (OR): Phase 2
Description: OR: confirmed stringent complete response(sCR),complete response(CR),very good partial response(VGPR) or partial response(PR) as per International Myeloma Working Group Uniform Response Criteria (IMWGURC). sCR: normal serum free light chain (FLC) ratio, absence of clonal cells in bone marrow. CR: disappearance of any soft tissue plasmacytomas, <5 percent (%) plasma cells in bone marrow, negative immunofixation on serum, urine. VGPR: serum, urine M-protein detectable by immunofixation but not on electrophoresis, >= 90% reduction in serum M-protein, <100 mg/24 hour (hr) urine M-protein. PR: >=50% reduction in serum M-protein, reduction in 24-hr urinary M-protein by >=90% or to <200 mg/24 hr, >=50% decrease in difference between involved and uninvolved FLC levels if serum, urine M-protein were unmeasurable, >= 50% reduction in plasma cells, provided baseline bone marrow plasma cell was >=30% if serum, urine M-protein were unmeasurable and serum free light assay was unmeasureable.
Time Frame: Cycle 1 Day 1 (baseline) up to end of study (up to cycle 22 for schedule B)
Population: Primary response analysis set (PRAS) included first consecutive (by first treatment day) participants in response analysis set (RAS=included all enrolled participants who received study treatment, had an adequate baseline tumor assessment and measurable disease) that were response-evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:ScheduleB)
Number analyzed (Participants) | 25
percentage of participants | 20 [6.8 to 40.7]

4. Secondary Outcome: Percent Change From Screening in Phosphorylated Retinoblastoma (Rb), Tumor Biomarkers and Soluble Biomarkers Levels: Phase 1
Time Frame: Screening, C1D1(baseline), C1D8, C1D15, C2D1, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1, C9D1, C10D1, C11D1, C12D1, C13D1, C14D1, C15D1, C16D1, C17D1, C18D1, C19D1, C20D1, C21D1, C22D1, End of Treatment (assessment at early withdrawal occurring up to Cycle 22)
Population: Results are not reported because data was present as individual participant listings but not summarized for analysis, as per change in planned analysis.
Groups:
- Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule A): Palbociclib (PD 0332991) 100 mg capsule orally once daily for 21 days followed by 7 days off-treatment in a 28-day cycle along with bortezomib 1.0 mg/m^2 intravenous injection and dexamethasone 20 mg tablet orally 30 minutes prior to bortezomib injection on Day 8, 11, 15 and 18 of 28-day cycle (schedule A) during Phase 1 of the study. Treatment was continued until any of the following withdrawal criteria was met: disease progression (unless the investigator judged that participant could still derive clinical benefit from continuing the treatment and the risk/benefit was still favorable), unacceptable toxicities, need for surgery or radiation therapy considered due to progressive disease by investigator, investigator conclusion that it is in the participant's best interest to discontinue therapy, need for anti-cancer therapy, lost to follow-up, withdrawal from treatment, or withdrawal of consent.
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule A) | Palbociclib 75mg+Bortezomib+Dexamethasone(Phase1:Schedule A) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule B) | Palbociclib 125mg+Bortezomib+Dexamethasone(Phase1:Schedule B)
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Best Overall Response: Phase 1
Description: Best overall response: best confirmed response on study after first study dose as per IMWGURC. sCR: normal FLC ratio, absence of clonal cells in bone marrow. CR: negative immunofixation on serum and urine, disappearance of any soft tissue plasmacytomas, <5% plasma cells in bone marrow. VGPR: serum and urine M-protein detectable by immunofixation but not on electrophoresis, >=90% reduction in serum M-protein, <100 mg/24 hr urine M-protein. PR: >=50% reduction of serum M-protein, reduction in 24-hr urinary M-protein by >=90% or to <200mg/24 hr. Progressive disease (PD): >=25% increase from lowest response level in serum M-component or urine M-component, >=10% bone marrow plasma cell percentage, definite development of new bone lesions/soft tissue plasmacytomas/definite increase in size of existing bone lesions/soft tissue plasmacytomas, development of hypercalcemia, attributed solely to plasma cell proliferative disorder. Stable disease (SD): criteria for CR, VGPR, PR or PD not met.
Time Frame: Cycle 1 Day 1 (baseline), assessed on Day 1 of every cycle up to end of study (up to Cycle 22 for schedule A and schedule B)
Population: RAS included all enrolled participants who received study treatment, had an adequate baseline tumor assessment and measurable disease.
Measure: Number; unit: participants
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule A) | Palbociclib 75mg+Bortezomib+Dexamethasone(Phase1:Schedule A) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule B) | Palbociclib 125mg+Bortezomib+Dexamethasone(Phase1:Schedule B)
Number analyzed (Participants) | 1 | 5 | 7 | 5
participants
  Stringent Complete Response | 0 | 0 | 0 | 0
  Complete Response | 0 | 0 | 0 | 0
  Very Good Partial Response | 0 | 1 | 0 | 1
  Partial Response | 0 | 0 | 0 | 0
  Stable Disease | 0 | 1 | 4 | 2
  Progressive Disease | 1 | 3 | 3 | 1
  Indeterminate | 0 | 0 | 0 | 1

6. Secondary Outcome: Time to Tumor Progression (TTP): Phase 2
Description: TTP was defined as the time from first dose of study medication to first documentation of objective tumor progression. TTP was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.44. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD] per IMWGURC). PD: >=25% increase from lowest response level in serum M-component or urine M-component, >=10% bone marrow plasma cell percentage, definite development of new bone lesions/soft tissue plasmacytomas/definite increase in size of existing bone lesions/soft tissue plasmacytomas, development of hypercalcemia, attributed solely to plasma cell proliferative disorder.
Time Frame: Cycle 1 Day 1 (baseline) up to 28 days after last dose of palbociclib
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:Schedule B): Palbociclib (PD 0332991) 100 mg capsule orally once daily for 12 days followed by 9 days off-treatment in a 21-day cycle along with bortezomib 1.0 mg/m^2 intravenous injection and dexamethasone 20 mg tablet orally 30 minutes prior to bortezomib injection on Day 8, 11, 15 and 18 of 21-day cycle (schedule B) during Phase 2 of the study. Treatment was continued until any of the following withdrawal criteria was met: disease progression (unless the investigator judged that participant could still derive clinical benefit from continuing the treatment and the risk/benefit was still favorable), unacceptable toxicities, need for surgery or radiation therapy considered due to progressive disease by investigator, investigator conclusion that it is in the participant's best interest to discontinue therapy, need for anti-cancer therapy, lost to follow-up, withdrawal from treatment, or withdrawal of consent.
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:Schedule B)
Number analyzed (Participants) | 30
months | 3.9 [1.4 to 7.4]

7. Secondary Outcome: Progression-free Survival (PFS): Phase 2
Description: PFS was the time from start of study treatment to date progressive disease was documented or death due to any cause, whichever occurred first. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.44. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death"). PD: >=25% increase from lowest response level in serum M-component or urine M-component, >=10% bone marrow plasma cell percentage, definite development of new bone lesions/soft tissue plasmacytomas/definite increase in size of existing bone lesions/soft tissue plasmacytomas, development of hypercalcemia, attributed solely to plasma cell proliferative disorder.
Time Frame: Cycle 1 Day 1 (baseline) up to 28 days after last dose of palbociclib
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:Schedule B)
Number analyzed (Participants) | 30
months | 3.9 [1.4 to 7.4]

8. Secondary Outcome: Duration of Objective Response (DR): Phase 2
Description: DR was defined as time from first documentation of objective tumor response (sCR, CR, VGPR or PR) that was subsequently confirmed to first documentation of objective tumor progression or death due to any cause since treatment started. sCR: normal FLC ratio, absence of clonal cells in bone marrow. CR: disappearance of any soft tissue plasmacytomas, <5% plasma cells in bone marrow, negative immunofixation on serum, urine. VGPR: serum, urine M-protein detectable by immunofixation but not on electrophoresis, >=90% reduction in serum M-protein, <100 mg/24hr urine M-protein. PR:>=50% reduction in serum M-protein, reduction in 24-hr urinary M-protein by >=90% or to <200 mg/24 hr. PD: >=25% increase from lowest response level in serum M-component, urine M-component, >=10% bone marrow plasma cell percentage, development of new bone lesions/soft tissue plasmacytomas/increase in size of existing bone lesions, development of hypercalcemia, attributed solely to plasma cell proliferative disorder.
Time Frame: Cycle 1 Day 1 (baseline) up to 28 days after last dose of palbociclib
Population: PRAS was defined as the first consecutive (by first treatment day) participants in RAS (RAS included all enrolled participants who received study treatment, had an adequate baseline tumor assessment and measurable disease) that were response-evaluable. DR was calculated for the subgroup of PRAS participants with objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:Schedule B)
Number analyzed (Participants) | 5
months | 4.63 [1.643 to NA] — Upper limit of 95% could not be estimated since very few number of participants had response.

9. Secondary Outcome: Overall Survival (OS): Phase 2
Description: OS was defined as the time from first dose of study medication to first documentation of death due to any cause. OS was calculated as (the death date or last known alive date [if death date unavailable] minus the date of first dose of study medication plus 1) divided by 30.44.
Time Frame: Cycle 1 Day 1 (baseline) up to end of study (up to Cycle 22 for schedule B), thereafter every 3 months until 1 year after the last dose of palbociclib
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:Schedule B)
Number analyzed (Participants) | 30
months | 21.1 [11.8 to NA] — Upper limit of confidence interval could not be estimated since majority of the participants were alive at the time of analysis.

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) by Severity: Phase 2
Description: An AE was any untoward medical occurrence attributed to study medication in a participant who received study medication. A serious AE (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Adverse events were graded according to the common terminology criteria for adverse events (CTCAE) criteria as 1=mild AE, 2=moderate AE, 3=severe AE, 4=life-threatening or disabling AE, 5=Death related to AE. The most severe grade was used in case of multiple occurrences of the same event.
Time Frame: Cycle 1 Day 1 (baseline) up to 28 days after last dose of palbociclib
Population: Safety analysis set (SAS) included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:Schedule B)
Number analyzed (Participants) | 30
participants
  Grade 2 | 2
  Grade 3 | 9
  Grade 4 | 18
  Grade 5 | 1

11. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Relationship to Study Medication: Phase 2
Description: An AE was any untoward medical occurrence attributed to study medication in a participant who received study medication. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study medication until 28 days after the last dose of study medication that were absent before treatment or that worsened relative to pretreatment state. All causality AEs included SAEs as well as non-serious AEs, without regard to relationship to the study medication, which occurred during the trial. Treatment-related were adverse events (serious as well as non-serious adverse events) considered related to study medication by the investigator. Number of participants with treatment related TEAEs and all causality TEAEs were summarized.
Time Frame: Cycle 1 Day 1 (baseline) up to 28 days after last dose of palbociclib
Population: SAS included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:Schedule B)
Number analyzed (Participants) | 30
participants
  All Causality | 30
  Treatment Related | 27

12. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Phase 2
Description: Laboratory parameters included hematology (hemoglobin, platelets, leukocytes, total neutrophils, eosinophils, basophils, lymphocytes, monocytes); liver function (total bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, albumin, total protein); renal function (creatinine, blood urea nitrogen, uric acid); electrolytes (sodium, potassium, chloride, bicarbonate, calcium, magnesium and phosphate); urinalysis (protein and immunology [C reactive protein]), and clinical chemistry (glucose). Total number of participants with laboratory abnormalities was reported.
Time Frame: Cycle 1 Day 1 (baseline) up to 28 days after last dose of palbociclib
Population: SAS included all enrolled participants who received at least 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:Schedule B)
Number analyzed (Participants) | 30
participants | 30

13. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30): Phase 2
Description: EORTC QLQ-C30: included functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting) and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea and financial difficulties). Most questions used 4 point scale (1 'Not at all' to 4 'Very much'); 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). Scores for functional scales, global health status and symptom scales were calculated as an average of individual items, transformed to 0-100 scale; higher score=better level of functioning, health status or greater degree of symptoms. Score of the single items were transformed to 0-100 scale; higher score=greater degree of symptom/difficulty.
Time Frame: C1D1 (baseline), C1D8, C1D15, C2D1, C3D1, C4D1, C5D1, C6D1, C7D1, C8D1, C9D1, C10D1, C11D1, C12D1, C13D1, C14D1, C15D1, C16D1, C17D1, C18D1, C19D1, C20D1, C21D1, C22D1, End of Treatment (assessment at early withdrawal occurring up to Cycle 22)
Population: Patient Reported Outcomes (PRO) analysis set included all enrolled participants who received study treatment, had a baseline PRO assessment, and completed at least 1 on-study PRO assessment. Here 'n' signifies those participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:Schedule B)
Number analyzed (Participants) | 27
units on a scale
  C1D1: Global Health Status (n=27) | 60.80 [50.7 to 70.9]
  C1D1: Physical Functioning (n=27) | 64.20 [55.6 to 72.8]
  C1D1: Role Functioning (n=27) | 59.88 [46.8 to 73.0]
  C1D1: Emotional Functioning (n=27) | 70.37 [59.8 to 80.9]
  C1D1: Cognitive Functioning (n=27) | 72.22 [62.0 to 82.4]
  C1D1: Social Functioning (n=27) | 69.14 [57.6 to 80.7]
  C1D1: Fatigue (n=27) | 29.63 [19.1 to 40.2]
  C1D1: Nausea and Vomiting (n=27) | 6.79 [2.2 to 11.4]
  C1D1: Pain (n=27) | 35.80 [22.0 to 49.6]
  C1D1: Dyspnea (n=27) | 32.10 [21.4 to 42.7]
  C1D1: Insomnia (n=27) | 43.21 [29.1 to 57.3]
  C1D1: Appetite Loss (n=27) | 20.99 [8.8 to 33.2]
  C1D1: Constipation (n=27) | 27.16 [12.5 to 41.8]
  C1D1: Diarrhea (n=27) | 11.11 [4.8 to 17.4]
  C1D1: Financial Problems (n=26) | 33.33 [17.2 to 49.5]
  C1D8: Global Health Status (n=26) | 60.58 [51.4 to 69.7]
  C1D8: Physical Functioning (n=26) | 67.18 [58.2 to 76.2]
  C1D8: Role Functioning (n=26) | 59.62 [47.0 to 72.3]
  C1D8: Emotional Functioning (n=26) | 72.76 [61.5 to 84.0]
  C1D8: Cognitive Functioning (n=26) | 69.87 [56.8 to 82.9]
  C1D8: Social Functioning (n=26) | 70.51 [58.3 to 82.8]
  C1D8: Fatigue (n=26) | 27.24 [16.0 to 38.5]
  C1D8: Nausea and Vomiting (n=26) | 12.82 [4.9 to 20.7]
  C1D8: Pain (n=26) | 42.31 [29.6 to 55.0]
  C1D8: Dyspnea (n=26) | 30.77 [18.2 to 43.4]
  C1D8: Insomnia (n=26) | 43.59 [29.0 to 58.2]
  C1D8: Appetite Loss (n=26) | 24.36 [10.3 to 38.4]
  C1D8: Constipation (n=26) | 34.62 [19.2 to 50.1]
  C1D8: Diarrhea (n=26) | 15.38 [5.1 to 25.6]
  C1D8: Financial Problems | 28.20 [15.2 to 41.2]
  C1D15: Global Health Status | 55.33 [45.2 to 65.5]
  C1D15: Physical Functioning (n=25) | 62.93 [54.1 to 71.7]
  C1D15: Role Functioning (n=25) | 52.67 [38.4 to 66.9]
  C1D15: Emotional Functioning (n=25) | 67.00 [55.2 to 78.8]
  C1D15: Cognitive Functioning (n=25) | 68.00 [56.8 to 79.2]
  C1D15: Social Functioning (n=25) | 64.00 [50.3 to 77.7]
  C1D15: Fatigue (n=25) | 33.00 [21.2 to 44.8]
  C1D15: Nausea and Vomiting (n=25) | 20.67 [10.5 to 30.8]
  C1D15: Pain (n=25) | 45.33 [32.7 to 58.0]
  C1D15: Dyspnea (n=25) | 42.67 [28.6 to 56.7]
  C1D15: Insomnia (n=25) | 40.00 [28.8 to 51.2]
  C1D15: Appetite Loss (n=25) | 29.33 [14.8 to 43.8]
  C1D15: Constipation (n=25) | 32.00 [16.9 to 47.1]
  C1D15: Diarrhea (n=25) | 20.00 [7.4 to 32.6]
  C1D15: Financial Problems (n=25) | 29.33 [16.0 to 42.7]
  C2D1: Global Health Status (n=25) | 52.33 [42.7 to 62.0]
  C2D1: Physical Functioning (n=25) | 63.73 [55.1 to 72.4]
  C2D1: Role Functioning (n=25) | 60.67 [50.2 to 71.2]
  C2D1: Emotional Functioning (n=25) | 65.67 [53.9 to 77.5]
  C2D1: Cognitive Functioning (n=25) | 72.00 [61.7 to 82.3]
  C2D1: Social Functioning (n=25) | 64.67 [52.5 to 76.8]
  C2D1: Fatigue (n=25) | 34.33 [22.5 to 46.1]
  C2D1: Nausea and Vomiting (n=25) | 12.67 [7.0 to 18.4]
  C2D1: Pain (n=25) | 43.33 [31.6 to 55.1]
  C2D1: Dyspnea (n=25) | 33.33 [22.8 to 43.8]
  C2D1: Insomnia (n=25) | 40.00 [28.1 to 51.9]
  C2D1: Appetite Loss (n=25) | 22.67 [9.7 to 35.7]
  C2D1: Constipation (n=25) | 21.33 [7.1 to 35.6]
  C2D1: Diarrhea (n=25) | 6.67 [1.0 to 12.3]
  C2D1: Financial Problems (n=25) | 29.33 [14.3 to 44.4]
  C3D1: Global Health Status (n=25) | 56.82 [48.1 to 65.5]
  C3D1: Physical Functioning (n=25) | 68.18 [59.2 to 77.2]
  C3D1: Role Functioning (n=22) | 62.88 [48.5 to 77.3]
  C3D1: Emotional Functioning (n=22) | 68.56 [56.5 to 80.6]
  C3D1: Cognitive Functioning (n=22) | 71.97 [59.8 to 84.1]
  C3D1: Social Functioning (n=22) | 70.45 [57.6 to 83.3]
  C3D1: Fatigue (n=22) | 31.44 [19.4 to 43.5]
  C3D1: Nausea and Vomiting (n=22) | 14.39 [5.5 to 23.3]
  C3D1: Pain (n=22) | 30.30 [16.7 to 43.9]
  C3D1: Dyspnea (n=22) | 36.36 [22.0 to 50.7]
  C3D1: Insomnia (n=22) | 36.36 [25.3 to 47.5]
  C3D1: Appetite Loss (n=22) | 22.73 [12.1 to 33.3]
  C3D1: Constipation (n=22) | 36.36 [22.0 to 50.7]
  C3D1: Diarrhea (n=22) | 6.06 [-1.3 to 13.5]
  C3D1: Financial Problems (n=22) | 34.85 [19.4 to 50.3]
  C4D1: Global Health Status (n=18) | 59.72 [49.6 to 69.8]
  C4D1: Physical Functioning (n=18) | 63.15 [51.0 to 75.3]
  C4D1: Role Functioning (n=18) | 60.19 [44.6 to 75.8]
  C4D1: Emotional Functioning (n=18) | 67.13 [53.8 to 80.5]
  C4D1: Cognitive Functioning (n=18) | 71.30 [57.7 to 84.9]
  C4D1: Social Functioning (n=18) | 64.81 [48.5 to 81.1]
  C4D1: Fatigue (n=18) | 32.87 [19.5 to 46.2]
  C4D1: Nausea and Vomiting (n=18) | 9.26 [2.2 to 16.4]
  C4D1: Pain (n=18) | 30.56 [16.8 to 44.3]
  C4D1: Dyspnea (n=18) | 37.04 [24.5 to 49.6]
  C4D1: Insomnia (n=18) | 35.19 [19.6 to 50.7]
  C4D1: Appetite Loss (n=18) | 20.37 [5.2 to 35.6]
  C4D1: Constipation (n=18) | 33.33 [17.3 to 49.4]
  C4D1: Diarrhea (n=18) | 5.56 [-3.0 to 14.1]
  C4D1: Financial Problems (n=18) | 33.33 [17.3 to 49.4]
  C5D1:Global Health Status (n=17) | 52.45 [42.2 to 62.7]
  C5D1: Physical Functioning (n=17) | 58.04 [47.1 to 69.0]
  C5D1: Role Functioning (n=17) | 56.86 [41.4 to 72.3]
  C5D1: Emotional Functioning (n=17) | 65.20 [49.5 to 80.9]
  C5D1: Cognitive Functioning (n=17) | 67.65 [52.1 to 83.2]
  C5D1: Social Functioning (n=17) | 59.80 [42.9 to 76.7]
  C5D1: Fatigue (n=17) | 34.80 [19.1 to 50.5]
  C5D1: Nausea and Vomiting (n=17) | 11.76 [4.5 to 19.0]
  C5D1: Pain (n=17) | 31.37 [16.3 to 46.5]
  C5D1: Dyspnea (n=17) | 45.10 [28.0 to 62.2]
  C5D1: Insomnia (n=17) | 27.45 [13.6 to 41.3]
  C5D1: Appetite Loss (n=17) | 17.65 [3.9 to 31.4]
  C5D1: Constipation (n=17) | 35.29 [18.7 to 51.9]
  C5D1: Diarrhea (n=17) | 9.80 [-3.4 to 23.0]
  C5D1: Financial Problems (n=17) | 27.45 [9.0 to 45.9]
  C6D1: Global Health Status (n=15) | 61.11 [50.8 to 71.4]
  C6D1: Physical Functioning (n=15) | 65.78 [55.6 to 75.9]
  C6D1: Role Functioning (n=15) | 61.11 [45.3 to 77.0]
  C6D1: Emotional Functioning (n=15) | 73.89 [59.1 to 88.7]
  C6D1: Cognitive Functioning (n=15) | 72.22 [56.0 to 88.5]
  C6D1: Social Functioning (n=15) | 71.11 [55.3 to 86.9]
  C6D1: Fatigue (n=15) | 26.11 [11.3 to 40.9]
  C6D1: Nausea and Vomiting (n=15) | 7.78 [0.1 to 15.5]
  C6D1: Pain (n=15) | 27.78 [14.9 to 40.7]
  C6D1: Dyspnea (n=15) | 31.11 [18.1 to 44.1]
  C6D1: Insomnia (n=15) | 31.11 [14.8 to 47.4]
  C6D1: Appetite Loss (n=15) | 11.11 [-4.0 to 26.2]
  C6D1: Constipation (n=15) | 28.89 [10.6 to 47.2]
  C6D1: Diarrhea (n=15) | 4.44 [-2.1 to 10.9]
  C6D1: Financial Problems (n=15) | 26.67 [9.3 to 44.0]
  C7D1: Global Health Status (n=11) | 53.79 [42.2 to 65.4]
  C7D1: Physical Functioning (n=11) | 56.36 [42.6 to 70.1]
  C7D1: Role Functioning (n=11) | 51.52 [27.8 to 75.2]
  C7D1: Emotional Functioning (n=11) | 66.67 [45.3 to 88.1]
  C7D1: Cognitive Functioning (n=11) | 74.24 [53.4 to 95.1]
  C7D1: Social Functioning (n=11) | 68.18 [46.1 to 90.3]
  C7D1: Fatigue (n=11) | 33.33 [11.9 to 54.7]
  C7D1: Nausea and Vomiting (n=11) | 12.12 [2.0 to 22.2]
  C7D1: Pain (n=11) | 37.88 [13.8 to 61.9]
  C7D1: Dyspnea (n=11) | 20.00 [3.3 to 36.7]
  C7D1: Insomnia (n=11) | 30.30 [9.2 to 51.4]
  C7D1: Appetite Loss (n=11) | 6.06 [-7.4 to 19.6]
  C7D1: Constipation (n=11) | 27.27 [7.7 to 46.8]
  C7D1: Diarrhea (n=11) | 12.12 [-3.0 to 27.2]
  C7D1: Financial Problems (n=11) | 27.27 [5.3 to 49.3]
  C8D1: Global Health Status (n=10) | 62.50 [48.7 to 76.3]
  C8D1: Physical Functioning (n=10) | 56.00 [39.0 to 73.0]
  C8D1: Role Functioning (n=10) | 58.33 [34.3 to 82.3]
  C8D1: Emotional Functioning (n=10) | 78.33 [65.4 to 91.3]
  C8D1: Cognitive Functioning (n=10) | 78.33 [60.5 to 96.1]
  C8D1: Social Functioning (n=10) | 73.33 [57.2 to 89.4]
  C8D1: Fatigue (n=10) | 21.67 [8.7 to 34.6]
  C8D1: Nausea and Vomiting (n=10) | 5.00 [-0.8 to 10.8]
  C8D1: Pain (n=10) | 31.67 [12.6 to 50.7]
  C8D1: Dyspnea (n=10) | 30.00 [6.3 to 53.7]
  C8D1: Insomnia (n=10) | 36.67 [10.4 to 62.9]
  C8D1: Appetite Loss (n=10) | 10.00 [-1.5 to 21.5]
  C8D1: Constipation (n=10) | 20.00 [-0.1 to 40.1]
  C8D1: Diarrhea (n=10) | 0.00 [0.0 to 0.0]
  C8D1: Financial Problems (n=10) | 40.00 [15.4 to 64.6]
  C9D1: Global Health Status (n=9) | 56.48 [41.5 to 71.4]
  C9D1: Physical Functioning (n=9) | 57.78 [39.5 to 76.1]
  C9D1: Role Functioning (n=9) | 68.52 [43.3 to 93.7]
  C9D1: Emotional Functioning (n=9) | 75.00 [62.2 to 87.8]
  C9D1: Cognitive Functioning (n=9) | 72.22 [49.1 to 95.3]
  C9D1: Social Functioning (n=9) | 74.07 [57.0 to 91.2]
  C9D1: Fatigue (n=9) | 25.00 [12.2 to 37.8]
  C9D1: Nausea and Vomiting (n=9) | 5.56 [-0.9 to 12.0]
  C9D1: Pain (n=9) | 25.92 [14.6 to 37.2]
  C9D1: Dyspnea (n=9) | 33.33 [11.1 to 55.5]
  C9D1: Insomnia (n=9) | 40.74 [19.4 to 62.1]
  C9D1: Appetite Loss (n=9) | 11.11 [-7.0 to 29.2]
  C9D1: Constipation (n=9) | 18.52 [-0.1 to 37.1]
  C9D1: Diarrhea (n=9) | 7.41 [-9.7 to 24.5]
  C9D1: Financial Problems (n=9) | 40.74 [12.7 to 68.7]
  C10D1: Global Health Status (n=6) | 52.78 [26.4 to 79.1]
  C10D1: Physical Functioning (n=6) | 52.22 [38.6 to 65.8]
  C10D1: Role Functioning (n=6) | 50.00 [18.7 to 81.3]
  C10D1: Emotional Functioning (n=6) | 70.83 [42.2 to 99.4]
  C10D1: Cognitive Functioning (n=6) | 75.00 [48.5 to 101.5]
  C10D1: Social Functioning (n=6) | 83.33 [61.2 to 105.5]
  C10D1: Fatigue (n=6) | 29.17 [0.6 to 57.8]
  C10D1: Nausea and Vomiting (n=6) | 2.78 [-4.4 to 9.9]
  C10D1: Pain (n=6) | 33.33 [14.2 to 52.5]
  C10D1: Dyspnea (n=6) | 33.33 [-10.9 to 77.6]
  C10D1: Insomnia (n=6) | 44.45 [15.9 to 73.0]
  C10D1: Appetite Loss (n=6) | 16.67 [-12.6 to 45.9]
  C10D1: Constipation (n=6) | 16.67 [-12.6 to 45.9]
  C10D1: Diarrhea (n=6) | 0.00 [0.0 to 0.0]
  C10D1: Financial Problems (n=6) | 38.89 [-12.6 to 90.4]
  C11D1: Global Health Status (n=5) | 61.67 [39.0 to 84.3]
  C11D1: Physical Functioning (n=5) | 54.67 [39.9 to 69.5]
  C11D1: Role Functioning (n=5) | 53.33 [26.3 to 80.3]
  C11D1: Emotional Functioning (n=5) | 65.00 [29.6 to 100.4]
  C11D1: Cognitive Functioning (n=5) | 73.33 [30.4 to 116.2]
  C11D1: Social Functioning (n=5) | 66.66 [37.4 to 95.9]
  C11D1: Fatigue (n=5) | 35.00 [-0.4 to 70.4]
  C11D1: Nausea and Vomiting (n=5) | 6.67 [-11.8 to 25.2]
  C11D1: Pain (n=5) | 30.00 [7.3 to 52.7]
  C11D1: Dyspnea (n=5) | 20.00 [-17.0 to 57.0]
  C11D1: Insomnia (n=5) | 40.00 [21.5 to 58.5]
  C11D1: Appetite Loss (n=5) | 13.33 [-9.3 to 36.0]
  C11D1: Constipation (n=5) | 13.33 [-23.7 to 50.4]
  C11D1: Diarrhea (n=5) | 6.67 [-11.8 to 25.2]
  C11D1: Financial Problems (n=5) | 26.67 [-18.7 to 72.0]
  C12D1: Global Health Status (n=15) | 45.00 [9.5 to 80.5]
  C12D1: Physical Functioning (n=15) | 52.00 [36.1 to 67.9]
  C12D1: Role Functioning (n=15) | 43.33 [8.7 to 78.0]
  C12D1: Emotional Functioning (n=15) | 63.33 [20.9 to 105.7]
  C12D1: Cognitive Functioning (n=15) | 70.00 [43.0 to 97.0]
  C12D1: Social Functioning (n=15) | 50.00 [24.7 to 75.3]
  C12D1: Fatigue (n=15) | 36.67 [-5.7 to 79.1]
  C12D1: Nausea and Vomiting (n=15) | 6.67 [-11.8 to 25.2]
  C12D1: Pain (n=15) | 43.33 [24.8 to 61.8]
  C12D1: Dyspnea (n=15) | 40.00 [-14.0 to 94.0]
  C12D1: Insomnia (n=15) | 33.33 [4.1 to 62.6]
  C12D1: Appetite Loss (n=15) | 26.67 [-8.0 to 61.3]
  C12D1: Constipation (n=15) | 6.67 [-11.8 to 25.2]
  C12D1: Diarrhea (n=15) | 13.33 [-9.3 to 36.0]
  C12D1: Financial Problems (n=15) | 46.67 [-0.5 to 93.9]
  C13D1: Global Health Status (n=6) | 54.17 [27.2 to 81.1]
  C13D1: Physical Functioning (n=6) | 53.34 [38.0 to 68.7]
  C13D1: Role Functioning (n=6) | 55.56 [19.4 to 91.7]
  C13D1: Emotional Functioning (n=6) | 69.44 [32.5 to 106.4]
  C13D1: Cognitive Functioning (n=6) | 69.44 [39.3 to 99.6]
  C13D1: Social Functioning (n=6) | 61.11 [34.8 to 87.4]
  C13D1: Fatigue (n=6) | 30.56 [-6.4 to 67.5]
  C13D1: Nausea and Vomiting (n=6) | 5.56 [-8.7 to 19.8]
  C13D1: Pain (n=6) | 27.78 [9.7 to 45.8]
  C13D1: Dyspnea (n=6) | 22.22 [-6.3 to 50.8]
  C13D1: Insomnia (n=6) | 27.78 [-6.6 to 62.2]
  C13D1: Appetite Loss (n=6) | 16.67 [-2.5 to 35.8]
  C13D1: Constipation (n=6) | 16.67 [-12.6 to 45.9]
  C13D1: Diarrhea (n=6) | 22.22 [-20.1 to 64.6]
  C13D1: Financial Problems (n=6) | 38.89 [-2.0 to 79.8]
  C14D1: Global Health Status (n=6) | 61.11 [43.9 to 78.3]
  C14D1: Physical Functioning (n=6) | 54.45 [40.9 to 68.0]
  C14D1: Role Functioning (n=6) | 50.00 [27.9 to 72.1]
  C14D1: Emotional Functioning (n=6) | 73.61 [45.7 to 101.5]
  C14D1: Cognitive Functioning (n=6) | 83.33 [61.2 to 105.5]
  C14D1: Social Functioning (n=6) | 69.45 [41.4 to 97.5]
  C14D1: Fatigue (n=6) | 26.39 [-1.5 to 54.3]
  C14D1: Nausea and Vomiting (n=6) | 2.78 [-4.4 to 9.9]
  C14D1: Pain (n=6) | 33.33 [14.2 to 52.5]
  C14D1: Dyspnea (n=6) | 22.22 [4.2 to 40.3]
  C14D1: Insomnia (n=6) | 22.22 [-6.3 to 50.8]
  C14D1: Appetite Loss (n=6) | 0.00 [0.0 to 0.0]
  C14D1: Constipation (n=6) | 16.67 [-12.6 to 45.9]
  C14D1: Diarrhea (n=6) | 5.56 [-8.7 to 19.8]
  C14D1: Financial Problems (n=6) | 33.33 [-10.9 to 77.6]
  C15D1: Global Health Status (n=6) | 66.67 [52.0 to 81.3]
  C15D1: Physical Functioning (n=6) | 52.23 [40.2 to 64.3]
  C15D1: Role Functioning (n=6) | 61.11 [34.8 to 87.4]
  C15D1: Emotional Functioning (n=6) | 61.11 [56.6 to 99.0]
  C15D1: Cognitive Functioning (n=6) | 72.22 [39.7 to 104.8]
  C15D1: Social Functioning (n=6) | 66.67 [35.4 to 98.0]
  C15D1: Fatigue (n=6) | 22.22 [1.0 to 43.4]
  C15D1: Nausea and Vomiting (n=6) | 2.78 [-4.4 to 9.9]
  C15D1: Pain (n=6) | 27.78 [3.9 to 51.7]
  C15D1: Dyspnea (n=6) | 27.78 [1.4 to 54.1]
  C15D1: Insomnia (n=6) | 22.22 [4.2 to 40.3]
  C15D1: Appetite Loss (n=6) | 5.56 [-8.7 to 19.8]
  C15D1: Constipation (n=6) | 16.67 [-12.6 to 45.9]
  C15D1: Diarrhea (n=6) | 5.56 [-8.7 to 19.8]
  C15D1: Financial Problems (n=6) | 44.45 [2.1 to 86.8]
  C16D1: Global Health Status (n=6) | 52.78 [28.9 to 76.7]
  C16D1: Physical Functioning (n=6) | 55.56 [46.0 to 65.1]
  C16D1: Role Functioning (n=6) | 50.00 [30.8 to 69.2]
  C16D1: Emotional Functioning (n=6) | 76.39 [47.4 to 105.4]
  C16D1: Cognitive Functioning (n=6) | 77.78 [56.6 to 99.0]
  C16D1: Social Functioning (n=6) | 69.44 [37.3 to 101.5]
  C16D1: Fatigue (n=6) | 23.61 [-5.4 to 52.6]
  C16D1: Nausea and Vomiting (n=6) | 0.00 [0.0 to 0.0]
  C16D1: Pain (n=6) | 33.33 [8.6 to 58.1]
  C16D1: Dyspnea (n=6) | 27.78 [1.4 to 54.1]
  C16D1: Insomnia (n=6) | 27.78 [1.4 to 54.1]
  C16D1: Appetite Loss (n=6) | 5.56 [-8.7 to 19.8]
  C16D1: Constipation (n=6) | 11.11 [-17.5 to 39.7]
  C16D1: Diarrhea (n=6) | 22.22 [-6.3 to 50.8]
  C16D1: Financial Problems (n=6) | 44.45 [2.1 to 86.8]
  C17D1: Global Health Status (n=6) | 55.56 [35.1 to 76.0]
  C17D1: Physical Functioning (n=6) | 51.11 [32.5 to 69.7]
  C17D1: Role Functioning (n=6) | 58.34 [43.7 to 73.0]
  C17D1: Emotional Functioning (n=6) | 73.61 [44.1 to 103.1]
  C17D1: Cognitive Functioning (n=6) | 72.22 [43.7 to 100.8]
  C17D1: Social Functioning (n=6) | 72.22 [45.9 to 98.6]
  C17D1: Fatigue (n=6) | 26.39 [-3.1 to 55.9]
  C17D1: Nausea and Vomiting (n=6) | 2.78 [-4.4 to 9.9]
  C17D1: Pain (n=6) | 30.56 [2.5 to 58.6]
  C17D1: Dyspnea (n=6) | 22.22 [-6.3 to 50.8]
  C17D1: Insomnia (n=6) | 50.00 [7.2 to 92.8]
  C17D1: Appetite Loss (n=6) | 5.56 [-8.7 to 19.8]
  C17D1: Constipation (n=6) | 22.22 [-13.9 to 58.4]
  C17D1: Diarrhea (n=6) | 5.56 [-8.7 to 19.8]
  C17D1: Financial Problems (n=6) | 44.45 [2.1 to 86.8]
  C18D1: Global Health Status (n=6) | 61.11 [43.9 to 78.3]
  C18D1: Physical Functioning (n=6) | 48.89 [37.5 to 60.3]
  C18D1: Role Functioning (n=6) | 50.00 [25.3 to 74.7]
  C18D1: Emotional Functioning (n=6) | 70.83 [34.7 to 107.0]
  C18D1: Cognitive Functioning (n=6) | 61.11 [18.7 to 103.5]
  C18D1: Social Functioning (n=6) | 63.89 [31.8 to 96.0]
  C18D1: Fatigue (n=6) | 29.17 [-7.0 to 65.3]
  C18D1: Nausea and Vomiting (n=6) | 8.33 [-13.1 to 29.8]
  C18D1: Pain (n=6) | 61.11 [25.0 to 97.2]
  C18D1: Dyspnea (n=6) | 33.33 [11.2 to 55.5]
  C18D1: Insomnia (n=6) | 33.33 [2.0 to 64.6]
  C18D1: Appetite Loss (n=6) | 22.22 [-6.3 to 50.8]
  C18D1: Constipation (n=6) | 22.22 [-13.9 to 58.4]
  C18D1: Diarrhea (n=6) | 5.56 [-8.7 to 19.8]
  C18D1: Financial Problems (n=6) | 44.44 [-3.4 to 92.2]
  C19D1: Global Health Status (n=4) | 45.83 [20.4 to 71.2]
  C19D1: Physical Functioning (n=4) | 45.00 [23.1 to 66.9]
  C19D1: Role Functioning (n=4) | 37.50 [-7.8 to 82.8]
  C19D1: Emotional Functioning (n=4) | 66.67 [9.4 to 124.0]
  C19D1: Cognitive Functioning (n=4) | 45.83 [-39.1 to 130.7]
  C19D1: Social Functioning (n=4) | 50.00 [12.5 to 87.5]
  C19D1: Fatigue (n=4) | 33.33 [-24.0 to 90.6]
  C19D1: Nausea and Vomiting (n=4) | 12.50 [-12.9 to 37.9]
  C19D1: Pain (n=4) | 58.33 [24.1 to 92.6]
  C19D1: Dyspnea (n=4) | 25.00 [-1.5 to 51.5]
  C19D1: Insomnia (n=4) | 41.67 [-25.1 to 108.4]
  C19D1: Appetite Loss (n=4) | 25.00 [-1.5 to 51.5]
  C19D1: Constipation (n=4) | 50.00 [-18.5 to 118.5]
  C19D1: Diarrhea (n=4) | 0.00 [0.0 to 0.0]
  C19D1: Financial Problems (n=4) | 41.67 [-25.1 to 108.4]
  C20D1: Global Health Status (n=2) | 37.50 [-15.5 to 90.5]
  C20D1: Physical Functioning (n=2) | 46.67 [-38.0 to 131.4]
  C20D1: Role Functioning (n=2) | 33.33 [33.3 to 33.4]
  C20D1: Emotional Functioning (n=2) | 33.33 [-284 to 351.0]
  C20D1: Cognitive Functioning (n=2) | 16.67 [16.6 to 16.7]
  C20D1: Social Functioning (n=2) | 41.67 [-64.2 to 147.6]
  C20D1: Fatigue (n=2) | 66.67 [-251 to 384.3]
  C20D1: Nausea and Vomiting (n=2) | 16.67 [-195 to 228.4]
  C20D1: Pain (n=2) | 66.67 [66.6 to 66.7]
  C20D1: Dyspnea (n=2) | 33.34 [-390 to 456.9]
  C20D1: Insomnia (n=2) | 50.00 [-162 to 261.8]
  C20D1: Appetite Loss (n=2) | 33.33 [33.3 to 33.4]
  C20D1: Constipation (n=2) | 16.67 [-195 to 228.4]
  C20D1: Diarrhea (n=2) | 16.67 [-195 to 228.4]
  C20D1: Financial Problems (n=2) | 83.34 [-128 to 295.1]
  C21D1: Global Health Status (n=1) | 41.67 [NA to NA] — 95% Confidence Interval (CI) was not estimable since only 1 participant was evaluable.
  C21D1: Physical Functioning (n=1) | 53.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Role Functioning (n=1) | 50.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Emotional Functioning (n=1) | 66.67 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Cognitive Functioning (n=1) | 0.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Social Functioning (n=1) | 33.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Fatigue (n=1) | 33.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Nausea and Vomiting (n=1) | 33.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Pain (n=1) | 66.67 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Dyspnea (n=1) | 0.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Insomnia (n=1) | 66.67 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Appetite Loss (n=1) | 33.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Constipation (n=1) | 0.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Diarrhea (n=1) | 0.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Financial Problems (n=1) | 100.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Global Health Status (n=1) | 16.67 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Physical Functioning (n=1) | 53.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Role Functioning (n=1) | 50.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Emotional Functioning (n=1) | 83.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Cognitive Functioning (n=1) | 33.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Social Functioning (n=1) | 33.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Fatigue (n=1) | 16.67 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Nausea and Vomiting (n=1) | 33.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Pain (n=1) | 83.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Dyspnea (n=1) | 0.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Insomnia (n=1) | 33.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Appetite Loss (n=1) | 0.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Constipation (n=1) | 0.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Diarrhea (n=1) | 0.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Financial Problems (n=1) | 100.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  End of treatment: Global health status (n=17) | 49.02 [34.7 to 63.4]
  End of Treatment: Physical Functioning (n=17) | 56.08 [45.0 to 67.2]
  End of Treatment: Role Functioning (n=17) | 56.86 [38.4 to 75.3]
  End of Treatment: Emotional Functioning (n=17) | 62.26 [49.1 to 75.4]
  End of Treatment: Cognitive Functioning (n=17) | 62.75 [48.7 to 76.8]
  End of Treatment: Social Functioning (n=17) | 65.69 [48.2 to 83.2]
  End of Treatment: Fatigue (n=17) | 37.74 [24.6 to 50.9]
  End of Treatment: Nausea and Vomiting (n=17) | 16.67 [4.5 to 28.8]
  End of Treatment: Pain (n=17) | 43.14 [26.0 to 60.3]
  End of Treatment: Dyspnea (n=17) | 41.18 [24.5 to 57.8]
  End of Treatment: Insomnia (n=17) | 49.02 [30.7 to 67.3]
  End of Treatment: Appetite Loss (n=17) | 25.49 [10.0 to 41.0]
  End of Treatment: Constipation (n=17) | 43.14 [27.4 to 58.9]
  End of Treatment: Diarrhea (n=17) | 5.88 [-3.2 to 14.9]
  End of Treatment: Financial Problems (n=17) | 45.10 [27.0 to 63.2]

14. Secondary Outcome: Quality of Life Questionnaire Multiple Myeloma Module (QLQ-MY20): Phase 2
Description: The QLQ-MY20 consisted of 20 items addressing 4 domains of health-related quality of life (HRQoL) important to participants with multiple myeloma: future perspective (2 items), pain/disease symptoms (6 items), social support /body image (2 items), and treatment side-effects (10 items). All items used 4 point scale (1 'Not at all' to 4 'Very much'). Scores for HRQoL domains were calculated as an average of the individual items, transformed to 0 to 100 range. Higher scores on symptom scales (disease symptoms and side effects of treatment) indicated a higher level of symptoms/problems. Higher scores on functional scales (future perspective and body image) indicated a higher level of QoL/functioning.
Time Frame: as for outcome 13
Population: PRO analysis set included all enrolled participants who received study treatment, had a baseline PRO assessment, and completed at least 1 on-study PRO assessment. Here 'n' signifies those participants who were evaluable at spefied time points for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:Schedule B)
Number analyzed (Participants) | 27
units on a scale
  C1D1: Disease Symptoms (n=27) | 35.68 [25.5 to 45.9]
  C1D1: Side Effects of Treatment (n=27) | 25.61 [17.7 to 33.5]
  C1D1: Future Perspective (n=27) | 46.50 [36.4 to 56.6]
  C1D1: Body Image (n=27) | 24.69 [11.2 to 38.2]
  C1D8: Disease Symptoms (n=25) | 35.51 [25.3 to 45.7]
  C1D8: Side Effects of Treatment (n=25) | 23.90 [16.1 to 31.7]
  C1D8: Future Perspective (n=25) | 44.44 [32.9 to 56.0]
  C1D8: Body Image (n=25) | 13.33 [3.6 to 23.1]
  C1D15: Disease Symptoms (n=25) | 32.31 [22.7 to 41.9]
  C1D15: Side Effects of Treatment (n=25) | 26.89 [19.8 to 33.9]
  C1D15: Future Perspective (n=25) | 48.89 [37.0 to 60.7]
  C1D15: Body Image (n=25) | 28.00 [14.4 to 41.6]
  C2D1: Disease Symptoms (n=25) | 29.82 [21.4 to 38.3]
  C2D1: Side Effects of Treatment (n=25) | 24.73 [18.5 to 31.0]
  C2D1: Future Perspective (n=25) | 46.22 [35.0 to 57.4]
  C2D1: Body Image (n=25) | 17.33 [7.5 to 27.2]
  C3D1: Disease Symptoms (n=21) | 25.13 [16.2 to 34.0]
  C3D1: Side Effects of Treatment (n=21) | 25.01 [18.1 to 31.9]
  C3D1: Future Perspective (n=21) | 44.44 [31.7 to 57.1]
  C3D1: Body Image (n=21) | 20.63 [10.5 to 30.8]
  C4D1: Disease Symptoms (n=18) | 28.71 [17.8 to 39.6]
  C4D1: Side Effects of Treatment (n=18) | 26.64 [18.0 to 35.3]
  C4D1: Future Perspective (n=18) | 44.45 [28.7 to 60.2]
  C4D1: Body Image (n=18) | 25.93 [8.4 to 43.5]
  C5D1: Disease Symptoms (n=17) | 27.78 [15.2 to 40.3]
  C5D1: Side Effects of Treatment (n=17) | 27.52 [19.1 to 36.0]
  C5D1: Future Perspective (n=17) | 45.75 [29.1 to 62.4]
  C5D1: Body Image (n=17) | 25.49 [11.2 to 39.7]
  C6D1: Disease Symptoms (n=15) | 24.08 [14.0 to 34.1]
  C6D1: Side Effects of Treatment (n=15) | 25.04 [15.2 to 34.9]
  C6D1: Future Perspective (n=15) | 40.74 [22.2 to 59.3]
  C6D1: Body Image (n=15) | 20.00 [1.8 to 38.2]
  C7D1: Disease Symptoms (n=11) | 25.96 [11.8 to 40.2]
  C7D1: Side Effects of Treatment (n=11) | 26.77 [11.5 to 42.0]
  C7D1: Future Perspective (n=11) | 44.44 [23.1 to 65.8]
  C7D1: Body Image (n=11) | 30.30 [9.2 to 51.4]
  C8D1: Disease Symptoms (n=10) | 18.56 [9.3 to 27.8]
  C8D1: Side Effects of Treatment (n=10) | 26.41 [9.8 to 43.0]
  C8D1: Future Perspective (n=10) | 35.56 [15.8 to 55.3]
  C8D1: Body Image (n=10) | 30.00 [9.1 to 50.9]
  C9D1: Disease Symptoms (n=9) | 19.14 [8.7 to 29.6]
  C9D1: Side Effects of Treatment (n=9) | 19.75 [10.8 to 28.7]
  C9D1: Future Perspective (n=9) | 39.51 [18.5 to 60.5]
  C9D1: Body Image (n=9) | 25.93 [4.6 to 47.3]
  C10D1: Disease Symptoms (n=6) | 25.93 [17.1 to 34.7]
  C10D1: Side Effects of Treatment (n=6) | 18.83 [5.9 to 31.7]
  C10D1: Future Perspective (n=6) | 33.33 [-4.3 to 70.9]
  C10D1: Body Image (n=6) | 16.67 [-12.6 to 45.9]
  C11D1: Disease Symptoms (n=6) | 18.52 [7.7 to 29.4]
  C11D1: Side Effects of Treatment (n=6) | 18.52 [7.3 to 29.8]
  C11D1: Future Perspective (n=6) | 38.89 [-4.6 to 82.4]
  C11D1: Body Image (n=6) | 22.22 [-6.3 to 50.8]
  C12D1: Disease Symptoms (n=5) | 28.89 [18.7 to 39.1]
  C12D1: Side Effects of Treatment (n=5) | 24.30 [8.1 to 40.5]
  C12D1: Future Perspective (n=5) | 53.33 [-2.2 to 108.9]
  C12D1: Body Image (n=5) | 40.00 [-14.0 to 94.0]
  C13D1: Disease Symptoms (n=6) | 25.00 [14.1 to 35.9]
  C13D1: Side Effects of Treatment (n=6) | 18.70 [5.4 to 32.0]
  C13D1: Future Perspective (n=6) | 37.04 [-5.8 to 79.8]
  C13D1: Body Image (n=6) | 33.33 [2.0 to 64.6]
  C14D1: Disease Symptoms (n=6) | 19.45 [11.4 to 27.5]
  C14D1: Side Effects of Treatment (n=6) | 18.64 [5.3 to 32.0]
  C14D1: Future Perspective (n=6) | 35.19 [-9.3 to 79.7]
  C14D1: Body Image (n=6) | 16.67 [-12.6 to 45.9]
  C15D1: Disease Symptoms (n=6) | 23.15 [6.9 to 39.4]
  C15D1: Side Effects of Treatment (n=6) | 18.09 [8.2 to 28.0]
  C15D1: Future Perspective (n=6) | 38.89 [-4.6 to 82.4]
  C15D1: Body Image (n=6) | 16.67 [-12.6 to 45.9]
  C16D1: Disease Symptoms (n=6) | 27.78 [9.3 to 46.2]
  C16D1: Side Effects of Treatment (n=6) | 16.91 [5.0 to 28.9]
  C16D1: Future Perspective (n=6) | 37.04 [-5.8 to 79.8]
  C16D1: Body Image (n=6) | 22.22 [-13.9 to 58.4]
  C17D1: Disease Symptoms (n=6) | 24.07 [11.0 to 37.2]
  C17D1: Side Effects of Treatment (n=6) | 19.26 [5.0 to 33.6]
  C17D1: Future Perspective (n=6) | 38.89 [-2.7 to 80.4]
  C17D1: Body Image (n=6) | 22.22 [-6.3 to 50.8]
  C18D1: Disease Symptoms (n=6) | 41.85 [25.9 to 57.8]
  C18D1: Side Effects of Treatment (n=6) | 18.52 [4.8 to 32.2]
  C18D1: Future Perspective (n=6) | 38.89 [-2.7 to 80.4]
  C18D1: Body Image (n=6) | 33.33 [2.0 to 64.6]
  C19D1: Disease Symptoms (n=4) | 43.06 [18.7 to 67.4]
  C19D1: Side Effects of Treatment (n=4) | 25.74 [4.6 to 46.8]
  C19D1: Future Perspective (n=4) | 38.89 [-29.6 to 107.4]
  C19D1: Body Image (n=4) | 41.67 [-25.1 to 108.4]
  C20D1: Disease Symptoms (n=2) | 44.45 [-96.8 to 185.7]
  C20D1: Side Effects of Treatment (n=2) | 35.19 [11.6 to 58.8]
  C20D1: Future Perspective (n=2) | 66.67 [-357 to 490.2]
  C20D1: Body Image (n=2) | 50.00 [-162 to 261.8]
  C21D1: Disease Symptoms (n=1) | 77.78 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Side Effects of Treatment (n=1) | 36.67 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Future Perspective (n=1) | 44.44 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C21D1: Body Image (n=1) | 33.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Disease Symptoms (n=1) | 61.11 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Side Effects of Treatment (n=1) | 33.33 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Future Perspective (n=1) | 44.44 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Body Image (n=1) | 66.67 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  End of Treatment: Disease Symptoms (n=17) | 37.58 [23.5 to 51.7]
  End of Treatment: Side Effects of Treatment (n=17) | 29.51 [21.5 to 37.6]
  End of Treatment: Future Perspective (n=17) | 46.41 [34.4 to 58.4]
  End of Treatment: Body Image (n=17) | 29.41 [13.5 to 45.3]

15. Secondary Outcome: Modified Version of Brief Pain Inventory - Short Form (m-BPI-sf) Questionnaire: Phase 2
Description: m-BPI-sf was a questionnaire designed to assess the severity of pain and the impact of pain on daily functions. m-BPI-sf contained questions that assessed pain severity (worst, least, average, right now) and pain interference (general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life). Each question was answered on a scale ranging from 0 "No pain" to 10 "Pain as bad as you can imagine". The 4 pain severity questions were averaged to derive an index of pain severity and the 7 function questions were averaged to derive an index for pain interference. Total score range for pain severity and interference indices: 0 to 10, where higher score indicated higher severity/interference.
Time Frame: as for outcome 13
Population: The PRO analysis set included all enrolled participants who received study treatment, had a baseline PRO assessment, and completed at least 1 on-study PRO assessment.'N' signifies those participants who were evaluable for this outcome measure and 'n' signifies participants who were evaluable at specified time points for each arm, respectively.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:Schedule B)
Number analyzed (Participants) | 26
units on a scale
  C1D1: Pain Severity (n=26) | 2.32 [1.4 to 3.2]
  C1D8: Pain Severity (n=25) | 2.62 [1.7 to 3.6]
  C1D15: Pain Severity (n=24) | 2.44 [1.5 to 3.4]
  C2D1: Pain Severity (n=24) | 2.30 [1.5 to 3.2]
  C3D1: Pain Severity (n=21) | 2.12 [1.2 to 3.1]
  C4D1: Pain Severity (n=17) | 2.02 [0.9 to 3.1]
  C5D1: Pain Severity (n=16) | 2.22 [1.0 to 3.4]
  C6D1: Pain Severity (n=14) | 1.66 [0.7 to 2.6]
  C7D1: Pain Severity (n=10) | 1.98 [0.5 to 3.5]
  C8D1: Pain Severity (n=9) | 2.47 [0.6 to 4.4]
  C9D1: Pain Severity (n=9) | 1.81 [0.5 to 3.1]
  C10D1: Pain Severity (n=6) | 1.08 [-0.1 to 2.3]
  C11D1: Pain Severity (n=5) | 1.45 [-0.0 to 2.9]
  C12D1: Pain Severity (n=5) | 1.67 [0.4 to 2.9]
  C13D1: Pain Severity (n=6) | 0.93 [0.1 to 1.7]
  C14D1: Pain Severity (n=6) | 1.42 [0.1 to 2.7]
  C15D1: Pain Severity (n=6) | 1.04 [-0.0 to 2.1]
  C16D1: Pain Severity (n=6) | 1.46 [0.0 to 2.9]
  C17D1: Pain Severity (n=6) | 1.67 [-0.3 to 3.6]
  C18D1: Pain Severity (n=6) | 2.88 [1.1 to 4.7]
  C19D1: Pain Severity (n=4) | 3.69 [1.3 to 6.1]
  C20D1: Pain Severity (n=2) | 3.50 [0.3 to 6.7]
  C21D1: Pain Severity (n=1) | 4.00 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Pain Severity (n=1) | 4.50 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  End of Treatment: Pain Severity (n=16) | 3.30 [1.9 to 4.6]
  C1D1: Pain Interference (n=25) | 2.53 [1.4 to 3.6]
  C1D8: Pain Interference (n=25) | 2.58 [1.4 to 3.7]
  C1D15: Pain Interference (n=23) | 3.06 [1.9 to 4.3]
  C2D1: Pain Interference (n=23) | 2.64 [1.5 to 3.7]
  C3D1: Pain Interference (n=21) | 2.34 [1.1 to 3.5]
  C4D1: Pain Interference (n=17) | 2.54 [1.2 to 3.9]
  C5D1: Pain Interference (n=16) | 2.74 [1.3 to 4.2]
  C6D1: Pain Interference (n=14) | 2.26 [0.8 to 3.7]
  C7D1: Pain Interference (n=10) | 2.94 [0.6 to 5.3]
  C8D1: Pain Interference (n=9) | 2.60 [0.6 to 4.6]
  C9D1: Pain Interference (n=9) | 2.13 [-0.0 to 4.3]
  C10D1: Pain Interference (n=6) | 2.07 [-0.1 to 4.2]
  C11D1: Pain Interference (n=5) | 2.40 [1.1 to 3.7]
  C12D1: Pain Interference (n=5) | 2.91 [1.0 to 4.8]
  C13D1: Pain Interference (n=6) | 1.90 [0.3 to 3.5]
  C14D1: Pain Interference (n=6) | 0.98 [-0.1 to 2.1]
  C15D1: Pain Interference (n=6) | 1.31 [0.2 to 2.4]
  C16D1: Pain Interference (n=6) | 1.83 [0.4 to 3.3]
  C17D1: Pain Interference (n=6) | 1.50 [0.4 to 2.6]
  C18D1: Pain Interference (n=6) | 2.86 [0.9 to 4.9]
  C19D1: Pain Interference (n=4) | 4.07 [2.1 to 6.0]
  C20D1: Pain Interference (n=2) | 5.07 [-14.0 to 24.1]
  C21D1: Pain Interference (n=1) | 2.57 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  C22D1: Pain Interference (n=1) | 6.71 [NA to NA] — 95% CI was not estimable since only 1 participant was evaluable.
  End of Treatment: Pain Interference (n=16) | 3.46 [1.9 to 5.0]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule A) | Palbociclib 75mg+Bortezomib+Dexamethasone(Phase1:Schedule A) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule B) | Palbociclib 125mg+Bortezomib+Dexamethasone(Phase1:Schedule B) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:ScheduleB)
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/6 | 0/7 | 5/5 | 10/30
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 7/7 | 5/5 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule A) (N=3) | Palbociclib 75mg+Bortezomib+Dexamethasone(Phase1:Schedule A) (N=6) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule B) (N=7) | Palbociclib 125mg+Bortezomib+Dexamethasone(Phase1:Schedule B) (N=5) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:ScheduleB) (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 2
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Central nervous system haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule A) (N=3) | Palbociclib 75mg+Bortezomib+Dexamethasone(Phase1:Schedule A) (N=6) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase1:Schedule B) (N=7) | Palbociclib 125mg+Bortezomib+Dexamethasone(Phase1:Schedule B) (N=5) | Palbociclib 100mg+Bortezomib+Dexamethasone(Phase2:ScheduleB) (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 1 | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 5
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 6 | 3 | 4 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 5 | 5 | 4 | 23
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 1 | 2
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 9
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 12
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 11
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 4
Tongue coated (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 3
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 6
Chills (General disorders) | 0 | 2 | 0 | 0 | 3
Fatigue (General disorders) | 1 | 1 | 2 | 2 | 21
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 3 | 8
Pain (General disorders) | 0 | 3 | 0 | 0 | 3
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 8
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 4
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood bicarbonate increased (Investigations) | 0 | 0 | 1 | 2 | 0
Blood bilirubin decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatinine decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 3 | 0 | 6
Blood glucose increased (Investigations) | 0 | 0 | 0 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 2 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 1 | 2 | 0
Blood potassium decreased (Investigations) | 0 | 1 | 1 | 1 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood sodium increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 1
Body height decreased (Investigations) | 0 | 1 | 0 | 0 | 0
General physical condition abnormal (Investigations) | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 2 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 0 | 3 | 2 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Overweight (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 2 | 9
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 8
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Coordination abnormal (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 6
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 8
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0 | 1
Hypogeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 1 | 1 | 9
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Renal injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Walking aid user (Social circumstances) | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 4
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Haemoglobinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 2
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 4
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gingival inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Palatal oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 1
Catheter site pruritus (General disorders) | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Spinal pain (General disorders) | 0 | 0 | 0 | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Meningitis pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1
Clostridium test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Granulocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 3
pH urine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Monoplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Listless (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.